CLINICAL TRIAL: NCT07213505
Title: Investigating New Front-end Features in the SONNET 3
Brief Title: This Clinical Investigation Assesses the Safety and Performance of a New Beamformer for MED-EL Cochlear Implant Recipients.
Acronym: M11S3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Collaborators: Medizinische Universität Innsbruck, Universitätsklinik für Hör-, Stimm-, und Sprachstörungen (Unknown); Universitätsklinikum St. Pölten - NÖ Landeskliniken, Universitätsklinikum für Hals-, Nasen-, Ohrenkrankheiten (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-EL_CRD_2024_01
Record Dates: First submitted 2025-08-25; First posted 2025-10-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cochlear Implant Users
Keywords: cochlear implant; audiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult MED-EL Cochlear implant users with post-lingual, severe to profound sensory-neural hearing los (Experimental): Testing new versus approved front-end features (within subject design)
  Interventions: Other: Testing new front-end features

INTERVENTIONS:
Other: Testing new front-end features — New front-end features (i,e, the Focused Beamformer which nhances directional hearing and the AI Mode Medium (utilizes adaptive intelligence for optimized sound processing) will be compared to the approved beamformer and AI mode) in a within subject design. Subjects will be fitted with a MED-EL SONNET 3 audio processor.

SUMMARY:
Cochlear implants help individuals with hearing loss by delivering electrical signals directly to the auditory nerve, bypassing damaged parts of the ear. While they significantly improve speech perception in quiet environments and over the telephone, challenges remain in noisy environments due to interference from background noise. To address this, advancements in signal-processing strategies, microphone technology, and noise-reduction algorithms have been introduced.

The focus of the study is on two new front-end features:

* Focused Beamformer - Enhances directional hearing.
* AI Mode Medium - Utilizes the adaptive intelligence for optimized sound processing.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of eighteen (18) years at time of enrolment
* Experienced MED-EL cochlear implant (CI) user (≥ 6 months) for the ear to be tested
* User of a MED-EL Audio Processor (i.e. a SONNET, SONNET 2, SONNET 3, or RONDO 3 ≥ 3months)
* Post-lingual onset of severe to profound sensory-neural hearing loss on the ear to be tested
* A minimum of 40% speech recognition in the Freiburg Monosyllables Test in quiet at 65 dB sound pressure level (SPL) for the ear to be tested (at the last time tested in clinical routine)
* Signed and dated Informed Consent Form (ICF) before the start of any study-specific procedure.

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* CI user with contralateral hearing equal to or better than 30 dB (pure-tone average over the following frequencies: 250, 500, 1000, and 2000 Hz)
* Implanted with C40X, or C40C on the ear to be tested
* Implanted with an auditory brainstem implant (ABI) or Split electrode array
* Known allergic reactions to components of the investigational medical device
* Anything that, in the opinion of the Investigator, would

  * place the subject at increased risk
  * preclude the subject's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Oldenburg Sentence Test in noise (S0 N±135) | immediately after the intervention
  Speech perception in noise measured in dB SNR (the new Focused beamformer and the Omnidirectional setting are tested)

SECONDARY OUTCOMES:
Oldenburg Sentence Test in noise (S0 N±135) | immediately after the intervention
  Speech perception in noise measured in dB SNR (the new Focused beamformer and the Natural beamformer are tested)
Oldenburg Sentence Test in noise (S0 N±135) | immediately after the intervention
  Speech perception in noise measured in dB SNR (theAI-Medium and the AI-Mild mode are tested)

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Medizinische Universität Innsbruck, Universitätsklinik für Hör-, Stimm-, und Sprachstörungen, Innsbruck
  - Universitätsklinikum St. Pölten, Abteilung für Hals-, Nasen- und Ohrenerkrankungen, Sankt Pölten

IPD SHARING:
Plan to Share IPD: No